CLINICAL TRIAL: NCT06419465
Title: Comparison of the Effects of Peer and Nurse Led Health Protection and Promotion Training Programs Based on Social Cognitive Theory on the Health Behaviors of Older People
Brief Title: The Effect of Health Protection and Promotion Training Programs on the Health Behavior of Older People
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Merve SIKLAROGLU, Research Assistant Merve SIKLAROGLU, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0286
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Older People; Health Promotion
Keywords: social cognitive theory; peer education; public health nursing; education; older people

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-Led Health Protection and Promotion Training Program (Experimental)
  Interventions: Behavioral: Peer-Led Health Protection and Promotion Training Program
- Health Protection and Promotion Training Program under the Leadership of a Public Health Nurse (Experimental)
  Interventions: Behavioral: Health Protection and Promotion Training Program under the Leadership of a Public Health Nurse

INTERVENTIONS:
Behavioral: Peer-Led Health Protection and Promotion Training Program — Multiple teaching methods will be used throughout 12 weeks; interactive group trainings on health protection and promotion issues and health seeking behavior methods, demonstration and demonstration using Google Fit and E-Nabiz mobile applications and downloading the applications to their phones, establishing WhatsApp groups to interact with peers, encouraging physical activity using the Google Fit mobile application. In order to provide social interaction, walking with peer leaders, health protection and development issues, receiving questions and opinions and giving guidance by individual phone calls regarding E-Nabiz and Google Fit mobile applications, holding peer group meetings and any of the Health Protection and Development Training Program targets. It consists of interventions such as giving a success badge for the relevant behavior if it reaches someone. Individual phone calls are also included in the intervention program.
  Arms: Peer-Led Health Protection and Promotion Training Program
Behavioral: Health Protection and Promotion Training Program under the Leadership of a Public Health Nurse — Multiple teaching methods will be used throughout 12 weeks; interactive group trainings on health protection and promotion issues and health seeking behavior methods, demonstration and demonstration using Google Fit and E-Nabiz mobile applications and downloading the applications to their phones, establishing WhatsApp groups to interact with nurses, encouraging physical activity using the Google Fit mobile application. To achieve any of the Health Protection and Development Training Program targets by walking with the nurse, taking individual phone calls regarding health protection and promotion issues, E-Nabiz and Google Fit mobile applications, receiving questions and opinions and giving guidance, holding group meetings in order to provide social interaction and social interaction. It consists of interventions such as giving a success badge for the relevant behavior. Individual phone calls are also included in the intervention program.
  Arms: Health Protection and Promotion Training Program under the Leadership of a Public Health Nurse

SUMMARY:
Protecting and improving health is an important intervention in preventing diseases, controlling chronic diseases and delaying their progression. Therefore, appropriate health promotion programs specific to elderly individuals need to be developed. Educational intervention is known to be effective in achieving behavioral change. This study differs from previous studies in that both peer (Intervention-1) and nurse-led (Intervention-2)-led education programs are planned as interventions. This research was designed as a mixed method study to compare the effects of Peer and Nurse Led Health Protection and Promotion Training Programs Based on Social Cognitive Theory (SCT) on the health behaviors of older people. The research will be carried out in two stages. The first phase was planned as a parallel two-arm non-randomized experimental study. This phase is planned to be carried out between November 2024 and January 2025 in two separate elderly homes in Muratpasa district of Antalya province, where older people are concentrated. The sample size was calculated as 108 older people (Intervention-1: 54, Intervention-2: 54). Intervention will be implemented for 12 weeks with the Health Protection and Promotion Training Program Based on SCT under peer leadership in the Intervention-1 group, and the same interventions will be carried out in the Intervention-2 group under the leadership of a nurse. Primary results of the research; health protection and promotion behavior practice, health promotion behavior practice level, self-efficacy belief and health seeking behavior. Secondary measurement results are; It is an assessment of blood pressure, blood sugar, body mass index and cardiovascular disease risk. Results will be measured before and 12 weeks after the intervention with the Health Protection and Promotion Behavior Checklist, Elderly Health Promotion Scale, General Self-Efficacy Scale, and Health Seeking Behavior Scale. In the second stage, it was planned to conduct two qualitative phenomenological design studies. In the first qualitative study, the investigators aimed to deeply understand the views of older people who received peer leader intervention and nurse intervention; In the second qualitative study, it was aimed to understand in depth the experiences of the older people as peer leaders in the health protection and promotion training program based on SCT. In the qualitative phase, the data will be based on the maximum diversity sampling method and will be collected through face-to-face in-depth individual interviews in the workshops of both elderly homes with Semi-Structured Interview Forms in February 2025.

ELIGIBILITY:
Inclusion Criteria:

* Low (for women: 0-4 points; for men: 0-3 points) or moderate (for women: 5-8 points; for men: 4-6 points) from the first part of the Health Protection and Promotion Behavior Checklist. Individuals aged 65 and over who score,
* Those who come to the elderly home where the research will be conducted at least once a week,
* Those residing in Antalya province,
* Those who have and can use a smartphone,
* Those who can speak and understand Turkish,
* Those who do not have dementia according to the Mini Mental State Assessment Test Short Form (those who score 9 points and above),
* Those who are independent according to the Katz Activities of Daily Living Scale (those who score 3 points and above),
* Those who agreed to participate in the study voluntarily,
* One elderly person from the same household will be included in this study.

Exclusion Criteria:

• Those who have previously received training on health protection will not be included in the research.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Health Protection and Promotion Behavior Checklist | Change in performing health protection and promotion behaviors and using E-Nabiz and Google Fit mobile applications at the twelfth week from baseline
  This form was prepared by researchers in line with the relevant literature in order to evaluate the health protection and promotion behaviors of individuals aged 65 and over and their use of E-Nabiz and Google Fit mobile applications. Health Protection and Promotion Behavior Checklist consists of three parts. The answers to this form will be evaluated as "Yes: 1 point", "No: 0 points". This form consists of low (for women: 0-14 points; for men: 0-13 points), medium (for women: 15-28 points; for men: 14-26 points) and high (for women: 29-42 points; For men: 27-40 points).
Elderly Health Promotion Scale | Change in the assessment of health promotion behaviors at the twelfth week from baseline
  It was developed to evaluate health-promoting behaviors in elderly individuals aged 65 and over and consists of 22 items and 6 subscales. On a four-point Likert-type scale, the elderly individual's responses to health promotion behavior implementation behaviors are; never (1 point), sometimes (2 points), often (3 points), always (4 points). Scores between 22 and 88 are obtained from the scale. Evaluation of the scale is done by summing the scores obtained from the questions belonging to each sub-dimension. A high score is interpreted as an increase in the frequency of the individual applying health-promoting behaviors belonging to the relevant sub-dimension.
General Self-Efficacy Scale | Change in general self-efficacy level at the twelfth week from baseline
  It was developed as 20 items to measure general self-efficacy and was revised by the same researchers in 1981, reducing the number of items to 10. The scale was prepared as a four-point Likert type, limited by completely false and completely true points. All items in the scale are scored positively, with a total score between 10 and 40. A high score means that general self-efficacy is high.
Health Seeking Behavior Scale | Change in health-seeking behavior at the twelfth week from baseline
  It consists of 12 items and 3 factors indicating health-seeking behavior. Health Search Behavior Scale covers online search behavior, professional search behavior and traditional search behavior factors. On a five-point Likert-type scale; The options are "1=I strongly disagree", "2=I disagree", "3=I am undecided", "4=I agree", "5=I strongly agree". The closer the averages obtained from the scale are to 5, the higher the health-seeking behavior, and the closer they are to 1, the lower the health-seeking behavior.

SECONDARY OUTCOMES:
Health Assessment Form | Change in the assessment of health at the twelfth week from baseline
  Health Evaluation Form; It consists of 27 questions that question blood pressure, blood sugar, body mass index (BMI) measurements and cardiovascular disease risk (CVD) assessment. The reason for making these measurements and evaluations in the Health Evaluation Form is the high incidence of hypertension, diabetes, obesity and CVD in the world and in Turkey, and these screenings are recommended for individuals aged 65 and over in the Guide to Periodic Examinations and Screening Tests Recommended in Family Medicine Practice. and active health screenings in the Disease Management Platform used in primary healthcare services.

IPD SHARING:
Plan to Share IPD: Undecided